CLINICAL TRIAL: NCT00829400
Title: Cognitive Training to Enhance VA Work Program Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDB0010-01101; D4752R (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2009-01-24; First posted 2009-01-27 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Mental Illness; Schizophrenia; Depression; PTSD; Bipolar Disorder
Keywords: Neuropsychology; Cognitive Remediation; Vocational Rehabilitation; Schizophrenia; Severe and persistent mental illness; Chronic and disabling mental illness
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Depression; Stress Disorders, Post-Traumatic; Bipolar Disorder; Bronchiolitis Obliterans Syndrome | interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posit Science (Experimental): Brain Fitness, Insight, and Aristotle Cognitive Software Training Suites Targeting 100 hours of training
  Interventions: Behavioral: Cognitive Remediation
- Nintendo Brain Age (Active Comparator): Brain Age 2 Nintendo DS Portable Device for home or office use, targeting 100 hours of training
  Interventions: Behavioral: Nintendo Brain Age

INTERVENTIONS:
Behavioral: Cognitive Remediation — Brain Fitness, Insight, and Aristotle Cognitive Remediation Software Suites Targeting 100 hours of training
  Other Names: Posit Science
  Arms: Posit Science
Behavioral: Nintendo Brain Age — Brain Age 2 Software Nintendo DS Portable for home or office use Targeting 100 hours of training
  Other Names: Nintendo
  Arms: Nintendo Brain Age

SUMMARY:
The purpose of this study is to determine whether augmenting work services with cognitive remediation can improve vocational outcomes for psychiatrically disabled participants in VA work services.

DETAILED DESCRIPTION:
Background: Our previous RR&D funded study demonstrated significantly better vocational outcomes for people with schizophrenia when cognitive training supplemented their participation in Incentive Therapy. We have found in a subsequent NIMH funded study involving cognitive training and supported employment that competitive employment outcomes were better for those who received cognitive training. Moreover, we found that patients with the poorest community function at intake were very unlikely to obtain competitive employment unless they received the cognitive training. The current study will test the effectiveness of cognitive training by extending it to a broader range of VA patients with psychotic disorders participating in all types of VA work services currently available, including Incentive Therapy, Compensated Work Therapy, and Supported Employment. We plan to offer it to any patient with a psychotic disorder who is unlikely to obtain competitive employment without additional services. We will also compare two types of cognitive training to determine whether cognitive game software works as well narrowly focused cognitive exercises.

Design and Method: This is a randomized clinical trial in which 80 VA patients referred for VA work services and who meet criteria for psychotic disorder and impaired community function will be randomized to one of two types of cognitive training. There will be two conditions with approximately 40 subjects per condition. Intake procedures will include psychosocial, neuropsychological, and psychiatric assessments. These assessments will be repeated at 6-months and 12 month follow-up. Cognitive training will consist of computer-based cognitive exercises of attention, memory and problem-solving and a weekly group that focuses on improving work behaviors. One of the computer-based systems employs engaging cognitive game software and the other uses specially designed exercises that narrowly focus on discrete cognitive processes. Work services will be provided as usual to both conditions. Primary endpoints are measures of productive activity including obtaining competitive employment, total hours worked, and money earned. Secondary endpoints include neuropsychological, quality of life and health status changes. The study will be for three years.

ELIGIBILITY:
Inclusion Criteria:

* Participant in VA work services
* Chronic and disabling psychiatric illness

Exclusion Criteria:

* Neurological Disease that may affect cognition
* Primary substance abuse
* Developmental Disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Work Activity | 6 month and 12 month

SECONDARY OUTCOMES:
Neuropsychological Assessment | 6 month and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Morris D Bell, PhD, Principal Investigator — VA RR&D, Yale University School of Medicine
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Background] Bell M, Bryson G, Greig T, Corcoran C, Wexler BE. Neurocognitive enhancement therapy with work therapy: effects on neuropsychological test performance. Arch Gen Psychiatry. 2001 Aug;58(8):763-8. doi: 10.1001/archpsyc.58.8.763. PMID 11483142
- [Background] Bell M, Fiszdon J, Greig T, Wexler B, Bryson G. Neurocognitive enhancement therapy with work therapy in schizophrenia: 6-month follow-up of neuropsychological performance. J Rehabil Res Dev. 2007;44(5):761-70. doi: 10.1682/jrrd.2007.02.0032. PMID 17943687
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Derived] Bell MD, Laws H, Pittman B, Johannesen JK. Comparison of focused cognitive training and portable "brain-games" on functional outcomes for vocational rehabilitation participants. Sci Rep. 2018 Jan 29;8(1):1779. doi: 10.1038/s41598-018-20094-w. PMID 29379114